CLINICAL TRIAL: NCT03015545
Title: The Effects of Whole Body Vibration (WBV) on Muscle Stiffness and Reflex Activity in People After Stroke.
Brief Title: The Effects of WBV on Muscle Stiffness and Reflex Activity in Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20161117007
Record Dates: First submitted 2016-12-29; First posted 2017-01-10 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Stroke
Keywords: Muscle Stiffness; Ultrasound elastography; H-reflex; Whole body vibration; blood perfusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This group will stand with knee flexion 60 degrees on the same vibration platform for 60 seconds for 5 times with 60-seconds rest interval, but no vibration will be given.
  Interventions: Device: paretic leg-control; Device: non-paretic leg-control
- High intensity whole body vibration (Active Comparator): This group will stand with knee flexion 60 degrees on the same vibration platform for 60 seconds for 5 times with 60-seconds rest interval. The whole body vibration platform will be set with frequency at 30Hz and amplitude at 1.5mm.
  Interventions: Device: paretic leg-WBV; Device: non-paretic leg-WBV

INTERVENTIONS:
Device: paretic leg-control — standing on the vibration platform, with no vibration signals delivered.
  Arms: Control
Device: paretic leg-WBV — standing on the vibration platform, with WBV at 30Hz, 1.5mm.
  Arms: High intensity whole body vibration
Device: non-paretic leg-control — standing on the vibration platform, with no vibration signals delivered.
  Arms: Control
Device: non-paretic leg-WBV — standing on the vibration platform, with WBV at 30Hz, 1.5mm.
  Arms: High intensity whole body vibration

SUMMARY:
Spastic hypertonia is common after stroke. Whole-body vibration (WBV) is known to have modulatory effects of muscle reflex activity and blood flow in other populations and thus have potential applications in the management of spastic hypertonia post-stroke. This study aims to investigate the acute effect of WBV on leg muscle H-reflex, stiffness, and blood perfusion in people with chronic stroke.

DETAILED DESCRIPTION:
Spastic hypertonia is common after stroke. Whole-body vibration (WBV) is known to have modulatory effects of muscle reflex activity and blood flow in other populations and thus have potential applications in management of spastic hypertonia post-stroke. However, the potential effects of WBV on leg muscle stiffness in stroke rehabilitation remains unknown. Scientific evidence is warranted to fill the knowledge gap.

Purpose This study aims to investigate the acute effect of WBV on leg muscle H-reflex, stiffness and blood perfusion in people with chronic stroke.

Methods Individuals with chronic stroke will be recruited from community self-help groups and existing patient database. Relevant information (e.g. demographic information, medical history) will be obtained from medical records and subject interviews. Each subject will have to fulfill the following inclusion criteria: (1) diagnosis of chronic stroke, (2) community-dwelling, (3) able to follow simple verbal instructions. Exclusion criteria are: (1) other diagnoses of neurological conditions, (2) significant musculoskeletal conditions (e.g. amputations), (3) metal implants in the lower extremity or spine, (4) recent fracture in the lower extremity, (5) diagnosis of osteoporosis, (6) vestibular disorders, (7) peripheral vascular disease, and (11) other serious illnesses or contraindications to exercise.

This is a single-blinded randomized within-patient cross-over study. Each participant was evaluated for the soleus H-reflex, stiffness and blood perfusion of the medial gastrocnemius (MG) using ultrasound on both sides before and after either a 5-minute WBV intervention (30 Hertz, 1.5mm, knee flexed 60 degrees) or a no-WBV condition (5 minutes). The measurements were performed at baseline and every 1-min post-intervention up to 5 minutes. The outcomes generated included the soleus H/M ratio, shear modulus and vascular index (VI) of the MG muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with a diagnosis of a hemispheric stroke >6 months,
2. Medically stable,
3. Able to stand independently for at least 1 minute and
4. Mas score >1 measured at the ankle plantar flexors.

Exclusion Criteria:

1. Brainstem or cerebellar stroke,
2. Other neurological condition,
3. Serious musculoskeletal or cardiovascular disease,
4. Severe contracture of the ankle that the cannot be put in the neutral position.
5. Metal implants or recent fractures in the lower extremities or spine,
6. Fresh skin wound in lower extremities, especially popliteal fossa
7. Other severe illnesses or contraindication for exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
H-reflex of paretic soleus muscle | Immediately before the intervention
  To measure the efficacy of synaptic transmission
H-reflex of paretic soleus muscle | 1st minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of paretic soleus muscle | 2nd minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of paretic soleus muscle | 3rd minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of paretic soleus muscle | 4th minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of paretic soleus muscle | 5th minute after the intervention
  To measure the efficacy of synaptic transmission
Muscle stiffness of paretic medial gastrocnemius | Immediately before the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of paretic medial gastrocnemius | 1st minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of paretic medial gastrocnemius | 2nd minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of paretic medial gastrocnemius | 3rd minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of paretic medial gastrocnemius | 4th minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of paretic medial gastrocnemius | 5th minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
H-reflex of non-paretic soleus muscle | Immediately before the intervention
  To measure the efficacy of synaptic transmission
H-reflex of non-paretic soleus muscle | 1st minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of non-paretic soleus muscle | 2nd minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of non-paretic soleus muscle | 3rd minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of non-paretic soleus muscle | 4th minute after the intervention
  To measure the efficacy of synaptic transmission
H-reflex of non-paretic soleus muscle | 5th minute after the intervention
  To measure the efficacy of synaptic transmission
Muscle stiffness of non-paretic medial gastrocnemius | Immediately before the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of non-paretic medial gastrocnemius | 1st minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of non-paretic medial gastrocnemius | 2nd minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of non-paretic medial gastrocnemius | 3th minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of non-paretic medial gastrocnemius | 4th minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position
Muscle stiffness of non-paretic medial gastrocnemius | 5th minute after the intervention
  Measured by Supersonic elastography with ankle in neutral position

SECONDARY OUTCOMES:
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | Immediately before the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | 1 minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | 2nd minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | 3rd minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | 4th minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of paretic medial gastrocnemius muscle | 5th minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of non-paretic medial gastrocnemius muscle | Immediately before the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of non-paretic medial gastrocnemius muscle | 1th minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of non-paretic medial gastrocnemius muscle | 2nd minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of non-paretic medial gastrocnemius muscle | 3rd minute after the intervention
  Measured by power Doppler ultrasound
MoviIntramuscular blood perfusion of non-paretic medial gastrocnemius muscle | 4th minute after the intervention
  Measured by power Doppler ultrasound
Intramuscular blood perfusion of non-paretic medial gastrocnemius muscle | 5th minute after the intervention
  Measured by power Doppler ultrasound

OTHER OUTCOMES:
Fugl-Meyer Assessment of Motor Recovery after Stroke--lower extremities | Immediately before the intervention
  Evaluates and measures motor recovery in post-stroke hemiplegic patients
Brief Balance Evaluation Systems Test | Immediately before the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hector WH Tsang, PhD, Study Chair — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No